CLINICAL TRIAL: NCT06324318
Title: A Multiregional RCT of Parenting in 2 Worlds for Urban American Indian Families
Brief Title: Parenting in 2 Worlds Multisite Trial
Acronym: (P2W)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Phoenix Indian Center (Unknown); Ain Dah Yung Center (Unknown); Denver Indian Center Inc (Unknown); Native American Community Services of Erie and Niagara Counties (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA056417 (NIH); R01DA056417 (NIH)
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Parenting; Mental Health Wellness 1; Substance Use; Risky Health Behavior
Keywords: family functioning; risky sexual behavior
MeSH Terms: conditions — Substance-Related Disorders; Health Risk Behaviors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parenting in 2 Worlds (treatment) (Experimental): A 10-week parenting intervention focused on improving overall family functioning and strengthen parenting skills to communicate with adolescents to avoid risk behaviors.
  Interventions: Behavioral: Parenting in 2 Worlds (P2W)
- Healthy Families in 2 Worlds (Active Comparator): A 10-week parenting intervention curriculum focused on improving parental knowledge of family health topics.
  Interventions: Behavioral: Healthy Families in 2 Worlds (HF2W)

INTERVENTIONS:
Behavioral: Parenting in 2 Worlds (P2W) — P2W is a culturally-adapted parenting intervention designed specifically for urban American Indian families. It is a 10-week, 10-lesson manualized curriculum with accompanying videos, designed to be facilitated by American Indians from the local communities. The workshop lessons cover topics like the identification of family values, culturally influenced child rearing values and traditions, sources of support for parents, and ways to improve parenting skills to communicate with, monitor, and guide adolescents to avoid substance use, unprotected sex and other risk behaviors
  Arms: Parenting in 2 Worlds (treatment)
Behavioral: Healthy Families in 2 Worlds (HF2W) — HF2W is a 10-week informational family health program. The workshop lessons cover topics such as oral health, CPR and first aid, dating safety, and teen mental health.
  Arms: Healthy Families in 2 Worlds

SUMMARY:
This research study will test the effectiveness of a culturally grounded parenting intervention called Parenting in 2 Worlds (P2W). This intervention is designed for American Indian / Alaska Native (AI) parents/guardians of adolescents who reside in urban areas. This will be a multi-regional effectiveness trial across four regions: Northeast (Buffalo/Niagara), Midwest (St. Paul/Minneapolis), Mountain (Denver), and Southwest (Phoenix). There are four specific aims. First, this study will test the effectiveness of Parenting in Two Worlds (P2W) as compared to an informational family health intervention, Healthy Families in 2 Worlds (HF2W), in improving parenting and family functioning. Second, this study will test if the relative effectiveness of P2W, compared to HF2W, varies by parent's/guardian's level of socioeconomic vulnerability, experiences of historical loss, or AI cultural identity. Third, this study will examine if P2W can reduce adolescent (ages 12 - 17) risky health behaviors including substance use, depressive symptoms, suicidality, and risky sexual behaviors. Fourth, this study will examine whether positive changes in parenting and family functioning that result from P2W lead to positive changes in adolescent's health behaviors.

DETAILED DESCRIPTION:
The study will conduct a comparative effectiveness trial, with a gender-stratified randomization of adults to alternate interventions in four urban communities. The overall objectives are to test the relative effectiveness of the culturally grounded Parenting in 2 Worlds (P2W) intervention for urban American Indian families in strengthening the proximal outcomes of family functioning and parenting skills, and distal outcomes in preventing adolescent risk behaviors. The investigators will employ Community-based Participatory Research approaches, with the participating urban Indian centers (UICs) partnering with the university research team and each other. Phase 1 has start-up, development, and planning activity, coordinated with a Community Advisory Board, to prepare the UICs to implement the intervention, develop capacity for recruiting, training, and program delivery. This process will integrally involve a UIC that has delivered P2W successfully (Phoenix Indian Center) to share its accumulated capacity-building and implementation expertise. American Indian workshop facilitators from the target communities will receive 2-day trainings on intervention delivery. In Phase 2, each UIC will first implement one cycle/round of the P2W intervention and the comparison group intervention, Healthy Families in 2 Worlds (HF2W) that served as a comparison group in the original Arizona efficacy trial of P2W. A facilitator for P2W and a facilitator for HF2W will each deliver their 10 weekly lessons, on a synchronized schedule. This first cycle will include pretest and post-test data collection and an on-going implementation process review to identify implementation challenges and solutions. After concluding the first cycle, project staff and facilitators from each UIC and the university research team will video conference to review successful implementation strategies and troubleshoot challenges. The UICs will then complete at least 5 additional cycles of delivering P2W and HF2W. For all cycles, each UIC will recruit American Indian parents or guardians of urban American Indian youth (aged 12-17) as workshop participants. Adult participants will be randomized individually, after stratification by gender, to receive the P2W or the HF2W curriculum. Both manualized curricula will be implemented at each site as originally designed, and surveys will be administered, in parallel time frames. Outcomes as reported by parents and by their designated adolescent child will be tracked over time through self-administered pretest and post-test questionnaires delivered on electronic platforms. Focus groups with parents will be conducted at each of the four study sites, after each of the two full implementation years, to provide insight into how P2W influenced their lives. An ongoing implementation review process will systematically record implementation decisions, challenges and solutions as identified by a range of stakeholders both within and across the four urban AI communities. Phase 3 will include data analysis and dissemination activities to community and academic audiences.

ELIGIBILITY:
Inclusion Criteria:

Adult participants:

* Must be American Indian parents or guardians of American Indian children aged 12 to 17 who attend urban schools
* Must reside in the service areas of the four urban Indian centers who are participating in this study
* Self-identifies as American Indian
* Must be primary caregiver responsible for day-to-day decisions for an American Indian child ages 12 to 17

Child Participants:

* Aged 12 - 17
* Identified by their parent/guardian as American Indian
* Attends an urban school

Exclusion Criteria:

* Not applicable

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in family functioning and cohesion | 10 week and 12 month follow up
  Caregiver and adolescent self-report about supportiveness, closeness, togetherness and cooperation among family members. Scale: Minimum = 1 and Maximum = 5 [1 = Almost never, 2 = Once in a while, 3 = Sometimes, 4 = Frequently, 5 = Almost always]. Higher is better outcome.
Change from baseline in parental involvement | 10 week and 12 month follow up
  Caregiver and adolescent self-report about caregiver's involvement in adolescent's daily activities. Scale: Minimum = 1 and Maximum = 4 [1 = More than 1 month ago, 2 = Within the last month, 3 = Within the last week, 4 = Yesterday or today]. Higher is better outcome.
Change from baseline in parental supervision | 10 week and 12 month follow up
  Caregiver and adolescent self-report about caregiver's direct supervision such as established curfews. Scale: Minimum = 1 and Maximum = 5 [1 = Almost never, 2 = Once in a while, 3 = Sometimes, 4 = Frequently, 5 = Almost always]. Higher is better outcome.
Change from baseline in parental monitoring | 10 week and 12 month follow up
  Caregiver and adolescent self-report about caregiver's knowledge of adolescent's activities, friends and whereabouts. Scale: Minimum = 1 and Maximum = 5 [1 = Almost never, 2 = Once in a while, 3 = Sometimes, 4 = Frequently, 5 = Almost always]. Higher is better outcome.
Change from baseline in positive parenting practices | 10 week and 12 month follow up
  Caregiver and adolescent self-report about caregiver's encouragement for good adolescent behavior. Scale: Minimum = 1 and Maximum = 5 [1 = Almost never, 2 = Once in a while, 3 = Sometimes, 4 = Frequently, 5 = Almost always]. Higher is better outcome.
Change from baseline in relational warmth | 10 week and 12 month follow up
  Caregiver self-report aspects of the parent-adolescent relationship like caring and responsiveness. Scale: Minimum = 1 and Maximum = 5 [1 = Almost never, 2 = Once in a while, 3 = Sometimes, 4 = Frequently, 5 = Almost always]. Higher is better outcome.
Change from baseline in relational hostility | 10 week and 12 month follow up
  Caregiver self-report aspects of the parent-adolescent relationship like anger, and demandingness. Scale: Minimum = 1 and Maximum = 5 [1 = Almost never, 2 = Once in a while, 3 = Sometimes, 4 = Frequently, 5 = Almost always]. Higher is worse outcome
Change from baseline in family conflict | 10 week and 12 month follow up
  Caregiver and adolescent self-report about positive and negative interactions in the parent-adolescent relationship. Scale: Minimum = 1 and Maximum = 5 [1 = Not at all, 2 = Only a little, 3 = Sometimes, 4 = Almost always, 5 = Almost]. Higher is worse outcome.
Change from baseline in parental self-agency | 10 week and 12 month follow up
  Caregiver self-reports on confidence in their ability to parent successfully and solve child rearing challenges. Scale: Minimum = 1 and Maximum = 5 [1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Very often, 5 = Always]. Higher is better outcome.
Change from baseline in effective discipline | 10 week and 12 month follow up
  Caregiver self-reports about difficulty in deciding and establishing effective rules and discipline for their adolescent. Scale: Minimum = 1 and Maximum = 6 [1 = Strongly disagree, 2 = Disagree, 3 = Disagree slightly, 4 = Agree slightly, 5 = Agree, 6 = Strongly agree]. Higher is better outcome.
Change from baseline in parental communication about sex | 10 week and 12 month follow up
  Caregiver self-reports about how open, responsive, and positive the communication is between parents and adolescents regarding safe sexual behaviors. Scale: Minimum = 1 and Maximum = 4 [1 =Never, 2 = A few times, 3 = Occasionally, 4 = Frequently]. Higher is better outcome.
Change from baseline in child problem behaviors. | 10 week and 12 month follow up
  Caregiver self-reports about their child's problem behaviors like being withdrawn/depressed, rule-breaking behavior, and aggressive behavior. Scale: Minimum = 0 and Maximum = 2 [0 = Not true, 1 = Somewhat or sometimes true, 2 =Very true or often true]. Higher is worse outcome.
Change from baseline in decision making about risk behaviors | 10 week and 12 month follow up
  Caregiver and adolescent self-report about both positive (e.g., leave the situation) and negative (e.g., react with anger) strategies they use to resist engaging in risk behaviors. Scale: Minimum = 0 and Maximum = 2 [0 = Never, 1 = Sometimes, 2 =Always. Higher is better outcome.
Change from baseline in substance use | 10 week and 12 month follow up
  Adolescent self-reports about their use of alcohol, tobacco, marijuana and other drugs in the past 30 days. Single items: Minimum = 0 and Maximum = 6 [0 = None, 1 = Once, 2 = 2-3 times, 3 = 4-9 times, 4 = 10-19 times, 5 = 20-39 times, 6 = 40 or more times]. Higher is better outcome.
Change from baseline in risky sexual behaviors | 10 week and 12 month follow up
  Adolescent self-reports about risky sexual behaviors like not using a condom or consuming alcohol before sexual intercourse. Single items: Minimum = 0 and Maximum = 1 [0 = No, 1 = Yes]. Higher is worse outcome.

SECONDARY OUTCOMES:
Change from baseline in depressive symptoms | 10 week and 12 month follow up
  Adolescent self-reports about their symptoms of depression like feeling sad. Scale: Minimum = 1 and Maximum = 4 [1 = Rarely or none of them time (less than 1 day), 2 = Some or a little of the time (1 - 2 days), 3 = Occasionally or a moderate amount of time (3 - 4 days), 4 = All of the time (5 - 7 days)]. Higher is worse outcome.
Change from baseline in suicidality | 10 week and 12 month follow up
  Adolescent self-reports about their suicidal ideation and behavior. Scale: Minimum = 0 and Maximum = 4 [0 = Never, 1 = Once, 2 = 1 - 2 times a week, 3 = 3 - 4 times a week, 4 = Daily]. Higher is worse outcome.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Phoenix Indian Center, Phoenix, Arizona
  - Denver Indian Center, Denver, Colorado
  - Ain Dah Yung Center, Saint Paul, Minnesota
  - Native American Community Services Erie and Niagara Counties, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No